CLINICAL TRIAL: NCT06713590
Title: A Phase 1, Open-Label, Randomized Study of Single-Dose Subcutaneous Axatilimab Compared With Intravenous Axatilimab in Healthy Participants
Brief Title: A Study to Evaluate a Single-Dose Subcutaneous Axatilimab Compared With Intravenous Axatilimab in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCA034176-102
Expanded Access: NCT05544032 (Available)
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Healthy Participants
Keywords: INCA34176; Axatilimab
MeSH Terms: interventions — axatilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental): Axatilimab will be administered at a protocol defined starting dose administered as an IV infusion.
  Interventions: Drug: Axatilimab
- Cohort B (Experimental): Axatilimab will be administered at a protocol defined starting dose administered as an SC injection.
  Interventions: Drug: Axatilimab
- Cohort C (Experimental): Axatilimab will be administered at a protocol defined starting dose administered as an SC injection.
  Interventions: Drug: Axatilimab
- Cohort D (Experimental): Axatilimab will be administered at a protocol defined starting dose administered as an SC injection.
  Interventions: Drug: Axatilimab

INTERVENTIONS:
Drug: Axatilimab — Axatilimab will be administered at protocol defined dose.

SUMMARY:
This study will be conducted to evaluate a Single-Dose Subcutaneous (SC) Axatilimab Compared With Intravenous Axatilimab in Healthy Participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Aged 18 to 55 years, inclusive, at the time of signing the ICF.
* Body mass index within the range of 18.0 to 30.0 kg/m2 (inclusive) at screening.

Note: Participants with a BMI up to 32.0 kg/m2 may be enrolled with the sponsor's approval.

* Body weight of ≥ 40 kg (inclusive). Note: For each cohort, approximately 6 participants from 1 of each weight band (40-65 kg, > 65-90 kg, > 90 kg) will be enrolled, to total approximately 24 participants in each weight band.
* No clinically significant findings on screening evaluations (clinical, ECG, and comprehensive physical examination, including the eyes). No laboratory values out of normal reference ranges.
* Ability to be administered IV or SC study drug.
* Willingness to avoid pregnancy or fathering children based on the protocol defined criteria below.

  * Male participants with reproductive potential must agree to take appropriate precautions to avoid fathering children, including refraining from donating sperm, from screening through 90 days (a spermatogenesis cycle) after the dose of study drug on Day 1 and must refrain from donating sperm during this period. Permitted methods in preventing pregnancy should be communicated to the participants and their understanding confirmed.
  * Female participants who are WOCBP must have a negative pregnancy test at screening and a negative pregnancy test at check-in (Day -1) and must agree to take appropriate precautions to avoid pregnancy from screening through 60 days (2 menstrual cycles) after the dose of study drug on Day 1 and must refrain from donating oocytes during this period. Permitted methods in preventing pregnancy should be communicated to the participants and their understanding confirmed.
  * Female participants not considered to be of childbearing potential as defined in the protocol are eligible and must have a negative pregnancy test at screening and check-in.

Exclusion Criteria:

* History of uncontrolled or unstable respiratory, renal, gastrointestinal, endocrine, hematopoietic, psychiatric, and/or neurological disease within 6 months of screening.
* History of cardiovascular, cerebrovascular, peripheral vascular, or thrombotic disease or uncontrolled hypertension.
* High blood pressure (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg at screening, confirmed by repeat testing).
* Resting pulse rate < 40 bpm or > 100 bpm at screening. May repeat up to 3 total measurements, separated by 5 minutes, to confirm.
* History of rheumatologic/autoimmune disorders, except for minor eczema and rosacea.
* History or presence of an abnormal ECG before initial dose administration that, in the investigator's opinion, is clinically significant. Participants with a QTcF interval > 470 milliseconds, regardless of sex. QRS interval > 120 milliseconds, or PR interval > 220 milliseconds will be excluded. In the event a value is exclusionary, a single ECG will be repeated twice, and an average taken of the 3 readings will be used to determine if a participant should be excluded.
* History of malignancy within 5 years of screening, with the exception of cured basal cell or squamous cell carcinoma of the skin, ductal carcinoma in situ, or Gleason 6 prostate cancer.
* Any major surgery within 4 weeks of screening.
* Donation of blood to a blood bank or participation in a clinical study (except a screening visit) within 4 weeks of screening (within 2 weeks for donation of plasma only).
* Blood transfusion within 4 months of check-in (Day -1).
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment (includes latent treated tuberculosis).
* Positive test for HBV, HCV, or HIV. Participants whose results are compatible with prior immunization for or immunity due to infection with HBV may be included at the discretion of the investigator.
* Any chronic or recurrent edema. History of urticaria, allergic rhinoconjunctivitis, seasonal atopic, food, and/or latex allergy.
* Medical or self-reported history of alcoholism within 3 months of screening.
* History of significant alcohol use within 3 months of screening, defined as regular alcohol consumption > 21 units per week for males and > 14 units for females (1 unit = one-half pint of beer or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine).
* Has received a live vaccine (including attenuated) or anticipation of need for such a vaccine during the study.

Note: No vaccines may be administered within 3 months prior to the first dose of study drug.

* Positive urine or breath test for ethanol or positive urine or serum screen for drugs of abuse that are not otherwise explained by permitted concomitant medications or diet.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug with another investigational medication or current enrollment in another investigational drug or investigational product study.
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity) deemed clinically relevant by the investigator.
* Previous receipt of axatilimab.
* Known hypersensitivity or severe reaction to axatilimab or excipients of axatilimab.
* Inadequate veins for multiple venous puncture or IV catheter insertion as determined by the investigator or designee.
* Inability or unlikeliness of the participant to comply with the dose schedule and study evaluations, in the opinion of the investigator.
* History of tobacco or nicotine-containing product use within 1 month of screening.
* Use of prescription drugs (including hormonal contraceptives) within 14 days of study drug administration or nonprescription medications/products (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days of study drug administration. However, occasional and standard-dose acetaminophen, ibuprofen, and standard-dose vitamins are permitted. Megadose vitamins or supplements are not permissible.
* Women who are pregnant or breastfeeding.
* Any condition that would, in the investigator's judgment: interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* eGFR < 90 mL/min/1.73 m2 based on the site's standard formula at screening. NOTE: assessment of eGFR may be repeated once if outside of the reference range.
* Excessive exercise beyond the activities of daily living (eg, Ironman®, triathlon, etc) within 7 days before check-in (Day -1).
* History of keloid or hypertrophic scarring.
* History of recurrent pneumonia, skin infection, or viral infections within 6 months of screening.
* History of acute or chronic pancreatitis.
* History of retinal eye disorders. Presbyopia, myopia, and astigmatism are permitted.
* Abdominal tattoos, scarring at injection site.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Parameter: Cmax of axatilimab | Pre dose and Post dose on Day 1, Post dose Days 2, 3, 4, 6, 8, 15, 22, 28 and 60
  Maximum Observed Plasma Concentration of axatilimab.
Pharmacokinetics Parameter: AUC(0-t) of axatilimab | Pre dose and Post dose on Day 1, Post dose Days 2, 3, 4, 6, 8, 15, 22, 28 and 60
  Area Under the concentration- time curve up to the last measurable concentration of axatilimab.
Pharmacokinetics Parameter: AUC 0-∞ of axatilimab | Pre dose and Post dose on Day 1, Post dose Days 2, 3, 4, 6, 8, 15, 22, 28 and 60
  Area Under the Concentration-time Curve From 0 to Infinity of axatilimab.
Number of participants with Treatment Emergent Advers Events (TEAE's) | Up to 3 months
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.

SECONDARY OUTCOMES:
ADA | Pre dose on Day 1, Post dose Days 8, 15, 22, 28 and 60
  Percent of patients with anti-drug antibody (ADA).
Pharmacokinetics Parameter: Tmax of axatilimab | Pre dose and Post dose on Day 1, Post dose Days 2, 3, 4, 6, 8, 15, 22, 28 and 60
  Time to reach maximum plasma concentration of axatilimab.
Pharmacokinetics Parameter: t1/2 of axatilima | Pre dose and Post dose on Day 1, Post dose Days 2, 3, 4, 6, 8, 15, 22, 28 and 60
  Apparent terminal phase disposition half-life of axatilimab.
Pharmacokinetics Parameter: CL (or CL/F) of axatilimab | Pre dose and Post dose on Day 1, Post dose Days 2, 3, 4, 6, 8, 15, 22, 28 and 60
  Dose clearance of axatilimab.
Pharmacokinetics Parameter: Vz (or Vz/F) of axatilimab | Pre dose and Post dose on Day 1, Post dose Days 2, 3, 4, 6, 8, 15, 22, 28 and 60
  Volume of distribution of axatilimab.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (1):
- Celerion, Inc, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Evaluate a Single-Dose Subcutaneous Axatilimab Compared With Intravenous Axatilimab in Healthy Participants — https://www.incyteclinicaltrials.com/study/?id=INCA034176-102&SearchTerm=INCA034176-102&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=